CLINICAL TRIAL: NCT07110532
Title: A Double-Blinded, Randomized Influenza Virus Challenge Trial of Recombinant Influenza RG-A/Arkansas/08/2020 (pH1N1) in Healthy Adults to Assess Safety and Optimal Infectious Dose
Brief Title: pH1N1 Blinded Challenge Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-0011; 75N93019C00055
Record Dates: First submitted 2025-07-17; First posted 2025-08-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-07-30

CONDITIONS: Influenza
Keywords: challenge; Double-blind; Influenza; Influenza A; pH1N1; Random
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Cohort 1A (Experimental): Subjects will randomly be administered a single intranasal virus (RG) -A/Arkansas/08/2020 (pH1N1) at a dose of 10^6 TCID50. One of the subjects will receive a sham dose of 0 TCID50. If the Protocol Safety Review Team (PSRT) agrees that the dose is safe then Cohort 1B and Cohort 2A will begin. If proven unsafe the dose will be de-escalated to Cohort XA. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort 1B (Experimental): Subjects will randomly be administered a single intranasal virus (RG) -A/Arkansas/08/2020 (pH1N1) at a dose of 10^6 TCID50. One of the subjects will receive a sham dose of 0 TCID50. If the PSRT agrees that the dose is safe then Cohort 1C and Cohort 2A will begin. If proven unsafe the dose will be de-escalated to Cohort XA. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort 1C (Experimental): Subjects will randomly be administered a single intranasal virus (RG) -A/Arkansas/08/2020 (pH1N1) at a dose of 10^6 TCID50. One of the subjects will receive a sham dose of 0 TCID50. If the PSRT agrees that the dose is safe then Cohort 2A will begin. If proven unsafe the dose will be de-escalated to Cohort XA. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort 2A (Experimental): Subjects will randomly be administered a single intranasal virus (RG) -A/Arkansas/08/2020 (pH1N1) at a dose of 10^7 TCID50. One of the subjects will receive a sham dose of 0 TCID50. If the PSRT agrees that the dose is safe then Cohort 2B will begin. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort 2B (Experimental): Subjects will randomly be administered a single intranasal virus, (RG) -A/Arkansas/08/2020 (pH1N1), at a dose of 10^7 TCID50. One of the subjects will receive a sham dose of 0 TCID50. If the PSRT agrees that the dose is safe then Cohort 2C will begin. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort 2C (Experimental): Subjects will randomly be administered a single intranasal virus, (RG) -A/Arkansas/08/2020 (pH1N1), at a dose of 10^7 TCID50. One of the subjects will receive a sham dose of 0 TCID50. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort XA (Experimental): Subjects will randomly be administered a single intranasal virus, (RG) -A/Arkansas/08/2020 (pH1N1), at a dose of 10^5 TCID50. One of the subjects will receive a sham dose of 0 TCID50. De-escalation will occur after PSRT review of Cohort 1A, Cohort 1B, and Cohort 1C. If the PSRT agrees that the dose is safe then Cohort XB will begin. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort XB (Experimental): Subjects will randomly be administered a single intranasal virus, (RG) -A/Arkansas/08/2020 (pH1N1), at a dose of 10^5 TCID50. One of the subjects will receive a sham dose of 0 TCID50. If the PSRT agrees that the dose is safe then Cohort XC will begin. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)
- Cohort XC (Experimental): Subjects will randomly be administered a single intranasal virus, (RG) -A/Arkansas/08/2020 (pH1N1), at a dose of 10^5 TCID50. One of the subjects will receive a sham dose of 0 TCID50. N=30
  Interventions: Biological: A/Arkansas/08/2020 (pH1N1); Other: Sham/Diluent (1X SPG+Arg+Gel)

INTERVENTIONS:
Biological: A/Arkansas/08/2020 (pH1N1) — GMP-grade, cell-based influenza A (pH1N1) virus (Lot #24-005), derived via reverse genetics for use in controlled human infection studies.
Other: Sham/Diluent (1X SPG+Arg+Gel) — Sterile diluent containing 1X Sucrose Phosphate Glutamate (SPG), 1% arginine, and 1% hydrolyzed gelatin, used as a sham comparator in the human challenge trial.

SUMMARY:
This protocol describes a clinical trial to develop and validate a Controlled Human Infection Model (CHIM) for influenza A/Arkansas/08/2020 (pH1N1). The study is designed to determine the optimal infectious dose of the pH1N1 challenge strain for use in future clinical trials evaluating influenza countermeasures. The study will enroll and challenge adult volunteers with the pH1N1 influenza virus challenge or sham inoculations. Given the adaptive design of this trial, the potential number of participants can vary. Depending on the pathway recommended by the PSRT and followed in the Trial Schema, the study population can range from around 30 to 120. However, it is anticipated that the final sample size will be around 60 participants receiving pH1N1 challenge product plus approximately 4 persons receiving a sham inoculation. Participants will be pre-screened for health and for serological HAI antibody titers of </1:40 against the challenge strain. Eligible participants will be enrolled sequentially into challenge cohorts and will be randomly assigned to receive a single dose of either sham inoculation or the interventional study product at a dose between 10^6 to 10^7 TCID50 (or 10^5 TCID50 if needed). Dose titration will be conducted under an adaptive escalation schedule whereby dosing will start at 10^6 TCID50 and escalate to the next dose if a pre-determined symptomatic influenza attack rate and clinical symptom score thresholds are not met and if the dose is determined to be safe with no pre-defined halting criteria being met.

The primary objectives of this study are to determine the optimal infectious dose of a pH1N1 viral challenge to cause laboratory-confirmed clinical influenza and to assess the safety profile of pH1N1 viral challenge.

DETAILED DESCRIPTION:
This protocol describes a clinical trial to develop and validate a Controlled Human Infection Model (CHIM) for influenza A/Arkansas/08/2020 (pH1N1). The study is designed to determine the optimal infectious dose of the pH1N1 challenge strain for use in future clinical trials evaluating influenza countermeasures. The study will enroll and challenge adult volunteers with the pH1N1 influenza virus challenge or sham inoculations. Given the adaptive design of this trial, the potential number of participants can vary. Depending on the pathway recommended by the PSRT and followed in the Trial Schema, the study population can range from around 30 to 120. However, it is anticipated that the final sample size will be around 60 participants receiving pH1N1 challenge product plus approximately 4 persons receiving a sham inoculation. Participants will be pre-screened for health and for serological HAI antibody titers of </=1:40 against the challenge strain. Eligible participants will be enrolled sequentially into challenge cohorts and will be randomly assigned to receive a single dose of either sham inoculation or the interventional study product at a dose between 10^6 to 10^7 TCID50 (or 10^5 TCID50 if needed). Dose titration will be conducted under an adaptive escalation schedule whereby dosing will start at 10^6 TCID50 and escalate to the next dose if a pre-determined symptomatic influenza attack rate and clinical symptom score thresholds are not met and if the dose is determined to be safe with no pre-defined halting criteria being met.

The primary objectives of this study are to determine the optimal infectious dose of a pH1N1 viral challenge to cause laboratory-confirmed clinical influenza and to assess the safety profile of pH1N1 viral challenge. The secondary objectives are to describe clinical symptoms following pH1N1 viral challenge, to describe viral detection by qualitative reverse transcription polymerase chain reaction (RT-PCR) and to describe the host serum influenza hemagglutination inhibition and microneutralization antibody responses.

ELIGIBILITY:
Inclusion Criteria:

1. Provides signed and dated informed consent form prior to the initiation of any trial procedures.
2. Able to understand and agrees to comply with all planned trial procedures and to be available for all study visits.
3. Age >/= 18 and </= 55 years at time of enrollment.
4. Must agree to collection of venous blood and nasal absorption specimens per protocol and enrollment in DMID 19-0025 biorepository protocol for use of residual/repository research blood specimens.
5. In good general health.*

   *Good health, as determined by medical history, medication use and physical examination to evaluate ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would not affect the assessment of the safety of participants or the immunogenicity of challenge. These medical diagnoses or conditions should be stable for the last 90 days -- no hospitalizations, emergency room or urgent care for condition (excluding musculoskeletal conditions). If a participant has an ongoing symptomatic condition for which they have had or have ongoing medical investigations but have not yet received a diagnosis or treatment plan, they may not be in good health, as determined by the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572. Participants may be on a medical intervention (such as device or medication) only if the condition or disease being treated is stable and not deteriorating, the medications are not listed in the Exclusion Criteria and treatment poses no additional risk to participant safety or assessment of adverse events. This also includes no change in prescription medication, dose, or frequency as a result of new symptoms or deterioration of the condition or disease being treated in the 30 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a condition or disease outcome (e.g., lowering of the dosage or frequency), as determined by the site Principal Investigator (PI) or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572, will not be considered a deviation of this inclusion criterion.
6. Able to take oral medication and willing to receive oseltamivir phosphate and/or baloxavir marboxil as part of the study.
7. Participants of childbearing potential* agree to the use of acceptable forms of contraception** for at least 30 days prior to enrollment and agree to use such a method during study participation.

   *Childbearing potential in a participant is defined as not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year since last menses if menopausal.

   **Acceptable forms of primary contraception include true abstinence (100% of time no insertional sexual intercourse), or, if heterosexual intercourse is anticipated, monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to enrollment, intrauterine devices, birth control pills, condoms, and injectable/implantable/insertable/transdermal hormonal birth control products. Must use at least one acceptable form of contraception for at least 30 days prior to enrollment and through study completion.
8. Non-smoker or non-habitual smoker* of tobacco, e-cigarettes, or marijuana

   *A non-habitual smoker is a person who smokes no more than four cigarettes, other tobacco products, e-cigarettes (to include vaping and Juul products), and/or marijuana in a week.
9. No self-reported or known history of alcoholism within the 2 years prior to enrollment.
10. No self-reported or known history of illicit drug use for at least 30 days prior to enrollment.
11. Agrees not to use the listed prescription or over the counter medications* within 7 days prior to confinement and through the confinement period**.

    *Oseltamivir, zanamivir, peramivir, baloxavir marboxil, amantadine, rimantadine, aspirin, intranasal steroids, decongestants, antihistamines, and non-steroidal anti-inflammatory drugs (NSAIDs)

    **An exception can be made with the approval of the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572
12. Screening pulse is 55 to 100 beats per minute, inclusive*

    *Screening pulse values in the normal range or with grade 1 abnormalities deemed not clinically significant by the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572 are considered acceptable.
13. Screening systolic blood pressure is 90 to 140 mmHg, inclusive*

    *Screening systolic blood pressure values in the normal range or with grade 1 abnormalities deemed not clinically significant by the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572 are considered acceptable.
14. Screening diastolic blood pressure is 55 to 90 mmHg, inclusive*

    *Screening diastolic blood pressure values in the normal range or with grade 1 abnormalities deemed not clinically significant by the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572 are considered acceptable.
15. Screening SpO2 >/= 95 percent
16. Screening respiratory rate is </= 16
17. Screening oral temperature is <100.4 degrees Fahrenheit
18. Screening body mass index (BMI) >/=18.5 and <40 kg/m^2 at screening 19 Screening
19. Screening lab test results are within acceptable parameters:*

    * White blood cell (WBC), Absolute lymphocyte count (ALC), Hemoglobin (Hgb), Platelet (PLT). Lab tests within normal range or with grade 1 abnormalities deemed not clinically significant by the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572 are considered acceptable.
    * Alanine transferase (ALT), Aspartate Aminotransferase (AST), Gamma-Glutamyl Transferase, Alkaline Phosphatase (ALP), Total Bilirubin, and Creatinine (Cr). Low values are acceptable for trial inclusion as they are not considered to be clinically significant.
20. Has a negative test result for hepatitis B surface antigen, hepatitis C virus antibody*, or HIV types 1 or 2 antibodies at screening.

    *Persons testing positive for hepatitis C virus antibody with a history of treatment and a negative HCV viral load may be acceptable in the opinion of the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572.
21. Electrocardiogram (ECG) and chest X-ray (CXR) at screening are within normal range or are not deemed clinically significant*

    *As determined by the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572.
22. Negative respiratory virus panel (including influenza A and B, and SARS-CoV-2) by certified polymerase chain reaction (PCR)-based assay on Day -2 and Day -1.
23. Agrees to remain in the confinement unit for at least 6 days after enrollment and until they meet discharge criteria.
24. Agrees to adhere to lifestyle considerations during the study. Note: Deviations of lifestyle considerations will be reported as protocol deviations but not as eligibility deviations.

Exclusion Criteria:

1. A history (self-reported or medically documented) of medical or psychiatric condition(s)* or physical exam finding that precludes participation.

   * Any condition that, in the opinion of the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572, might interfere with the safety of the participant and/or study objectives including, but not limited to the following:
   * Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications (Inhaled, oral, or intravenous corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics) or any treatment for respiratory disease exacerbations (e.g., asthma exacerbation) within the last 5 years
   * Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult
   * Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, encephalopathy, Guillain-Barre syndrome, encephalomyelitis, or transverse myelitis). A history of febrile seizures during childhood alone is not diagnostic of epilepsy.
   * Anatomic or neurologic abnormality impairing the gag reflex or contributing to aspiration
   * Significant abnormality altering anatomy of nose/nasopharynx (including significant nasal polyps), clinically significant nasal deviation, nasal/sinus surgery within 180 days prior to enrollment, spontaneous epistaxis requiring medical care within 180 days prior to enrollment, chronic or recurrent sinusitis (four or more distinct episodes of sinusitis, with symptom-free intervals between episodes) in the last year prior to enrollment
   * Significant immunodeficiency
   * Known infection by human immunodeficiency virus (HIV) or hepatitis B virus, or known untreated hepatitis C virus infection
   * Ongoing malignancy or diagnosis of malignancy in the last five years (excluding squamous cell or basal cell carcinoma of the skin)
   * Diabetes
   * Blood dyscrasias or significant disorder of coagulation
2. HAI antibody titer >1:40 against influenza A/Arkansas/08/2020 (pH1N1) at screening
3. Current or within 4-month use of medications that may be associated with impaired immune responsiveness* *Including, but not limited to, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids (i.e., exceeding 14 days of use and/or exceeding 10 mg/ day prednisone equivalent) or other similar or toxic drugs during the preceding 3-month period prior to screening. Low dose systemic corticosteroids (10mg/day or lower of prednisone) for 14 days or fewer are permitted. Low dose topical and intranasal steroid preparations are allowed, if not within 7 days of challenge or during the confinement period.
4. Current pregnancy* or lactation

   *Participants of childbearing potential must have a negative serum pregnancy test at screening, a negative urine pregnancy test after admission to the confinement unit but before challenge, and a negative pregnancy test before any CXR (if >/= 7 days have passed since a serum pregnancy test).
5. Presence of an internal cardiac device such as a pacemaker or other implanted electronic medical devices
6. Has received blood or blood products in the last six months or has plans to donate blood or blood products in the duration of the study
7. History of a previous severe allergic reaction to any drug or biologic with generalized urticaria, angioedema, or anaphylaxis
8. Allergy or intolerance to treatments for influenza (including any neuraminidase inhibitors or baloxavir marboxil)
9. Allergy to two or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides)
10. Allergy to excipients in the challenge virus inoculum
11. Presence of any febrile illness or symptoms suggestive of a respiratory infection at the time of enrollment, the time of confinement, or Day 1 pre-challenge
12. Close contact with anyone known or suspected to have a respiratory viral illness within 7 days prior to enrollment
13. Currently enrolled in any other investigational study or plans to enroll in any other study within the period of this study*

    *Co-enrollment in an observational study, an investigational study in a follow-up/post vaccination stage, or a study involving a licensed drug or biologic may be allowed at the discretion of the site PI or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572.
14. Received any live vaccine in the 4 weeks prior to enrollment.
15. Received any influenza vaccine in the 4 months prior to enrollment or plans to receive influenza vaccine during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants reporting a related SAE at any time from challenge. | Through Day 57
Number and percentage of participants reporting any related AE from challenge. | Through Day 29
Number and percentage of participants with symptomatic influenza virus infection. | Day 2 through Day 6
  "Symptomatic influenza virus infection" is defined as meeting both of these criteria:
  1. Viral shedding detected in NP swab specimens by qualitative RT-PCR; and
  2. A cumulative symptom score >/=6 using a Modified Jackson Score.
Number of related adverse events (AE) reported from challenge. | Through Day 29
Number of related serious adverse events (SAE) from challenge. | Through Day 57

SECONDARY OUTCOMES:
Duration of viral shedding quantified by number of days of qualitative RT-PCR influenza detections in NP swab samples | Through Day 6
  Using qualitative RT-PCR by dose and study day
Geometric Mean Fold Rise (GMFR). | Day 6 through 29
Geometric Mean Titers (GMTs). | Day 6 through 29
HAI and MN antibody geometric mean titers (GMTs) at baseline. | Before Day 0
Investigator-assessed clinical symptoms as measured by Modified Jackson Score, post challenge through antiviral administration. | Through Day 6
  By dose, qualitative RT-PCR detection status, and clinical case definition status
Investigator-assessed clinical symptoms as measured by Modified Jackson Score, post challenge. | Through Day 15
  By dose, qualitative RT-PCR detection status, and clinical case definition status
Number and percentage of participants with seroconversion by dose. | Day 6 through 29
Percentage of participants with influenza virus detected in nasopharyngeal (NP) swab sample. | Through Day 6
  Using quantitative RT-PCR by dose
Self-reported clinical symptoms as measured by FLU-PRO/Validation Diary, post challenge through antiviral administration. | Through Day 6
  By dose, qualitative RT-PCR detection status, and clinical case definition status
Self-reported clinical symptoms as measured by FLU-PRO/Validation Diary, post challenge. | Through Day 15
  By dose, qualitative RT-PCR detection status, and clinical case definition status

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Duke Vaccine and Trials Unit, Durham, North Carolina